CLINICAL TRIAL: NCT00299442
Title: Can Self-Help Parent Training Reduce Conduct Problems in Children on NHS Waiting Lists for Child Mental Health Services?
Brief Title: Self-Help Parent Training for Conduct Problems in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Dr. Paul Montgomery, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/Q1606/57; ISRCTN12814243
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2008-11

CONDITIONS: Behavioral Symptoms
Keywords: behavior; conduct; child; parenting; self-help; media-based
MeSH Terms: conditions — Behavioral Symptoms; Behavior | interventions — (tris(diphenylphosphinomethyl)phenylborate)(p-tolylnitrido)iron(I)

ARMS (2):
- 1 (Experimental): Self-help Triple P Behavioural Family Intervention
  Interventions: Behavioral: Self-help Triple P Behavioural Family Intervention
- 2 (No Intervention): Wait-list control

INTERVENTIONS:
Behavioral: Self-help Triple P Behavioural Family Intervention — 10-week self-help workbook and videos
  Other Names: Triple P
  Arms: 1

SUMMARY:
This project will introduce a self-help parent training programme for families on National Health Service (NHS) waiting lists for child mental health services. It will examine whether access to treatment can be increased by providing an intervention that requires fewer resources and by releasing clinician time for more serious cases. This intervention will be tested in a randomised, controlled trial in which 35 subjects will receive treatment immediately and 35 will receive treatment after waiting for 10 weeks. All families will also complete questionnaires before and after the 10 week study period in order to measure changes in child behaviour, parenting, and parental mental health. Cost-effectiveness of this programme will also be analysed. Intention-to-treat analyses will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Families on waiting lists and child and adolescent mental health services clinics with children aged 2-5.
* Scores in the clinical range on a standardised measure of child behaviour problems.
* At least one parent in each family must be literate, fluent English speakers to participate because the self-administered intervention will primarily consist of written instructions and information in English.

Exclusion Criteria:

* Clients whose children score below a clinical cut-off score on a standardised measure of child behaviour problems. This is to ensure that participants are appropriate for an intervention aiming to reduce behaviour problems.
* Non-English speakers or those who are unable to read cannot be included because reading English is required to complete the self-administered intervention.
* Children or parents with severe disabilities and children with a developmental disorder (e.g., autism) will be excluded because the version of the parent training programme that will be implemented is not designed for families with these types of problems.
* Children who live with a temporary caregiver will be excluded because the intervention is designed for full-time parents and follow-up will be after one year.
* Children or parents who are currently receiving treatment for psychological problems will be excluded because outcomes may be influenced by interventions not affiliated with this project.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-02 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Eyberg Child Behavior Inventory | 6 months
Sutter-Eyberg Student Behavior Inventory | 10 weeks
Parent Daily Report | 6 months

SECONDARY OUTCOMES:
Depression-Anxiety Stress Scale | 10 weeks
Parent Sense of Competence Scale | 10 weeks
Parenting Scale | 10 weeks
Dyadic Adjustment Scale | 10 weeks
Strengths and Difficulties Questionnaire | 10 weeks
Therapy Attitude Inventory | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Montgomery, D. Phil., Principal Investigator — University of Oxford
Locations (3):
- United Kingdom (3):
  - West Berkshire PCT, Reading, Berkshire
  - Wycombe CAMHS, High Wycombe, Buckinghamshire
  - Sue Nicholls Centre, Aylesbury, Bucks

REFERENCES:
- [Background] Montgomery P, Bjornstad G, Dennis J. Media-based behavioural treatments for behavioural problems in children. Cochrane Database Syst Rev. 2006 Jan 25;2006(1):CD002206. doi: 10.1002/14651858.CD002206.pub3. PMID 16437442